CLINICAL TRIAL: NCT03808961
Title: NAPS: Niacin for Parkinson's Disease
Brief Title: Low Dose Niacin (Vitamin B3) for Parkinson's Disease
Acronym: NAPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough recruitment
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: NURE-013-18S
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease, Niacin, Niacinamide; Niacin; Niacinamide
MeSH Terms: conditions — Parkinson Disease | interventions — Niacin; Niacinamide

STUDY DESIGN:
Intervention Model Description: There are three arms, niacin, niacinamide and placebo. They are double blind and randomized.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only Pharmacists keep the log of the drug dispensed. Everyone else is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 - Niacin Arm (Active Comparator): Oral 100 mg fixed dose twice daily x 18-months (200 mg total / day) with assessments @ baseline, 6 month, 12 month and 18 months
  Interventions: Dietary Supplement: Niacin
- Group 2 - Niacinamide Arm (Active Comparator): Oral 100 mg fixed dose twice daily (200 mg total / day) x 18-months with assessments @ baseline, 6 month, 12 month and 18 months
  Interventions: Dietary Supplement: Niacinamide
- Group 3 - Placebo Wait-listed Arm (Placebo Comparator): Oral placebo twice daily x 18- months with assessments @ baseline, 6 month, 12 month and 18 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Niacin — 100mg tablets twice daily
  Other Names: Vitamin B3, Nicotinic acid
  Arms: Group 1 - Niacin Arm
Dietary Supplement: Niacinamide — 100mg tablets twice daily
  Other Names: Vitamin B3, Nicotinamide
  Arms: Group 2 - Niacinamide Arm
Other: Placebo — Placebo tablet twice daily
  Arms: Group 3 - Placebo Wait-listed Arm

SUMMARY:
(1) To examine the blood, urine and spinal fluid of persons with Parkinson's to look for evidence of inflammation and; (2) whether 18 months of vitamin B3(niacin or niacinamide) supplementation may reduce the inflammation and/or improve PD motor and non-motor symptoms.

DETAILED DESCRIPTION:
Number of people affected by Parkinson's disease is increasing each year. Vitamin B3 (Niacin/Niacinamide) supplement can be used to slow the progression of PD.

Inflammation plays a central role in Parkinson's disease (PD) pathology as evidenced by the presence of microglia in the substantia nigra in post-mortem samples as well as activated microglia and cytokines in clinical and animal studies. The use of non-aspirin non-steroidal anti-inflammatory drugs was found to reduce the risk of PD. The investigators recently identified an anti-inflammatory receptor GPR109A that is upregulated in PD. Niacin has a high affinity for this receptor, suggesting that it (niacin) may play an important role in reducing inflammation in PD. The investigators also found that individuals with PD have a chronic niacin deficiency. In a three month trial at Augusta University (the investigators' affiliate) the investigators demonstrated that niacin was helpful for PD patients in reducing inflammatory macrophages and boosting the anti-inflammatory macrophages in blood.

In this VA-funded study, the investigators will determine the effect of 18 months over-the-counter (OTC) niacin or niacinamide supplementation on inflammation (as assessed in the blood and spinal fluid) and severity of the PD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* PD subjects will be adult men and women diagnosed with idiopathic mild to moderately severe PD
* The majority of PD subjects are expected to be > 60 years old
* Disease severity is defined as modified Hoehn & Yahr Stages I-IV (while "On")
* PD is defined according to the UK Brain Bank Criteria made at least six months prior to recruitment to the study
* PD features include the presence of at least two of the four cardinal clinical manifestations of the disease, which are:

  * tremor
  * rigidity
  * bradykinesia
  * disturbances of posture or gait, without any other known or suspected cause of Parkinsonism
* Subjects should be stabilized on PD medication for at least 3 months before enrollment into the study
* Subjects' PD drug prescriptions will not be altered nor withheld during the study
* The patient will have signed informed consent

Exclusion Criteria:

* Subjects will be excluded if they present with significant cognitive deficits
* A MMSE score of 25 is considered substantial global cognitive impairment
* Subjects will be excluded if they had previous brain surgery or other severe neurological problems

  * intracerebral hemorrhage
  * traumatic brain injury
  * central nervous system malignancy
  * active central nervous system (CNS) infection
  * significant stroke
  * Alzheimer disease or any type of implanted stimulator including but not limited to Deep Brain Stimulator (DBS) or pacemaker
* All subjects must be without evidence of dementia

  * defined as a score > 24 the Mini-Mental State Examination and able to understand test instructions
* Subjects must not have functional blindness (inability to participate in gait and visuomotor assessments) or lower limb amputation higher than the forefoot or any orthopedic problem that precludes performance of physical tests
* Subjects must not have known allergy to vitamin B3
* Significant cardiac, pulmonary, hepatic, gastrointestinal, renal disease, or uncontrolled/advanced diabetes are also exclusionary factors, e.g.:

  * New York Heart Association Class III or IV congestive heart failure
  * endocarditis
  * pulmonary insufficiency symptomatic at rest or with mild physical exertion
  * acute or chronic hepatitis
  * renal failure requiring dialysis
  * second and third degree atrioventricular (AV) block
  * sick sinus syndrome
* Subjects will be excluded if they are taking B3 but will be included if they are taking B complex that has very low dose B3 (25 mg) which has minimal effects on GPR109A (based on our unpublished observation)
* Overall, the investigators will exercise clinical judgment to exclude a subject from the study if, in the investigators' opinion, that a patient presents with a set of comorbidities which renders unsuitability for the study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandramohan Wakade, MBBS, Principal Investigator — Charlie Norwood VA Medical Center, Augusta, GA
Locations (1):
- Charlie Norwood VA Medical Center, Augusta, GA, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
At the investigators request, we will share the data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after the study is closed.
Access Criteria: When we are ready to publish, the data will be available

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 - Niacin Arm | Group 2 - Niacinamide Arm | Group 3 - Placebo Wait-listed Arm
Started | 2 | 2 | 3
Completed | 2 | 2 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Al participants were tested for mini mental exam, UPDRS III, Visual analogue fatigue scale, 15 feet step score, and a trail making scores.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Niacin Arm | Group 2 - Niacinamide Arm | Group 3 - Placebo Wait-listed Arm | Total
Number analyzed (Participants) | 2 | 2 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 0 | 2
  >=65 years | 1 | 1 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8) | 67.5 (3.5) | 69.33 (2.5) | 66.27 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 1 | 2 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 1 | 2 | 2 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 3 | 7
UPDRS III [Mean (Standard Deviation); unit: units on a scale.] — UPDRS III score ranges from 0-132. Lower the score, better the outcome.
  units on a scale. | 40.5 (9) | 20.5 (4) | 17.6 (8) | 26.2 (12)
Mini Mental examination [Mean (Standard Deviation); unit: units on a scale] — Mini Mental score ranges from 0-30. Higher scores denote better outcome. Scores below 23 are excluded from study because they have major cognitive issues.
  units on a scale | 30 (0) | 28.5 (2.5) | 30 (0) | 29.5 (0.5)
Visual Analogue Fatigue Score [Mean (Standard Deviation); unit: score on a scale] — It is a self-assessed subjective score. It ranges from 0-10. 0 = no fatigue and 10 =major fatigue.
  score on a scale | 6.5 (0.5) | 5.5 (0.5) | 7 (3) | 6.3 (1.2)
step score [Mean (Standard Deviation); unit: seconds] — The subject is asked to walk 15 steps in one direction, turn back and walk 15 steps again. The noted time is in seconds to complete 15 steps.
  seconds | 20.4 (0.4) | 13 (2) | 10.4 (2.2) | 14.6 (4)
Trail making [Mean (Standard Deviation); unit: seconds] — Trail making test A comprises of tracing numbers sequentially and test B consists of alternating between tracing a number and an alphabet, starting from 1 and A. Lower scores in seconds demonstrate better hand-eye coordination and better cognitive function.
  seconds
    A | 35.5 (5.5) | 72.5 (31.5) | 49.33 (21) | 52.44 (18.69)
    B | 81.5 (9) | 150.5 (65.5) | 198 (203.22) | 143.33 (58.57)

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Change
Description: This is the Unified Parkinson's disease rating scale assessment. The investigators assess part III of the UPDRS regarding motor skills. The values reported are the averages of baseline, 6months, 12 months, and 18 months values combined for all the participants in that group. So, in the niacin and the niacinamide groups, it indicated the average of 8 values and in the control group it is the average of 12 values. A score is recorded according to the motor skills recorded ranging from 0-5 in each test, 0 being normal and 5 being affected most. Scores are given judging the motor skills. The score may range between 0-132. Lower scores indicate better outcome.
Time Frame: Baseline, 6 month, 12 month and 18 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 - Niacin Arm | Group 2 - Niacinamide Arm | Group 3 - Placebo Wait-listed Arm
Number analyzed (Participants) | 2 | 2 | 3
score on a scale | 40.5 (10) | 20.5 (2.5) | 17.5 (12)

2. Primary Outcome: Mini-Mental State Examination (MMSE) Change
Description: It captures mental status and awareness of time, place and surrounding. Score ranges from 0-30, 30 denotes the best score and best mental status. All the values in the group are pooled for an average score at baseline, 6 months, 12 months, and 18 months. Therefore, Niacin and Niacinamide groups each demonstrates average of 8 values while placebo group shows average of 12 values.
Time Frame: Baseline, 6 month, 12 month and 18 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 - Niacin Arm | Group 2 - Niacinamide Arm | Group 3 - Placebo Wait-listed Arm
Number analyzed (Participants) | 2 | 2 | 3
score on a scale | 29.57 (1.04) | 29.4 (1.2) | 30 (0)

3. Secondary Outcome: Visual Analogue Fatigue Scale Changes
Description: Fatigue is self-reported on the Visual analogue fatigue scale (VAFS). Participants were asked about how much fatigue they feel ranging from no fatigue (score 0) to extreme fatigue (score 10). Each participant was asked about this score at baseline, 6 months, 12 months, and 18 months visit. Data reported is the averages of all the scores from that group for all the time points.
Time Frame: Baseline, 6 month, 12 month and 18 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 - Niacin Arm | Group 2 - Niacinamide Arm | Group 3 - Placebo Wait-listed Arm
Number analyzed (Participants) | 2 | 2 | 3
score on a scale | 5.75 (1.5) | 5.75 (1.5) | 8.8 (2.5)

4. Secondary Outcome: Trail Making Test Time Change
Description: This is a timed test where the patient connects numbers in order for part A. Numbers and letters are connected interchangeably in past B. The time of B minus the time of A gives a measure for set shift change ability which is reduced in Parkinson's patients. Each A and B demonstrates averages from baseline, 6 months, 12 months and 18 months of all the participants. Therefore, in the niacin group A and group B each show averages of 8 values while the control group shows averages of 12 values.
Time Frame: Baseline, 6 month, 12 month and 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months
Description: Any event after taking the medication such as allergies, redness, difficulty in breathing etc.
Arm/Group | Group 1 - Niacin Arm | Group 2 - Niacinamide Arm | Group 3 - Placebo Wait-listed Arm
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT03808961/Prot_SAP_000.pdf